CLINICAL TRIAL: NCT01062945
Title: The Effects of Doxazosin on the Cardiovascular and Subjective Effects of Cocaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas Newton, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-25442; P50DA018197 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Cocaine Addiction; Cocaine Abuse; Cocaine Dependence; Substance Abuse
Keywords: Cocaine; Doxazosin
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Sugars; Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Doxazosin (Active Comparator)
  Interventions: Drug: Doxazosin

INTERVENTIONS:
Drug: Placebo — Matching administration of a placebo pill.
  Other Names: Sugar pill
  Arms: Placebo
Drug: Doxazosin — The dose of doxazosin needed to alter the effects of cocaine is unknown and preclinical animal studies have not been conducted. Because of this, initially we will study the effects of a low dose of doxazosin (4 mg daily) compared to placebo daily. Because this class of medication needs to be titrated upward due to the potential for hypotension, treatment will begin at 1 mg and increased by 1 mg increments every three days until 4 mg is reached on day 12.
  Other Names: Cardura
  Arms: Doxazosin

SUMMARY:
The purpose of the study is to asses the potential interactions between intravenous cocaine and doxazosin in cocaine dependent volunteers who are not seeking treatment. The study will evaluate the effects of doxazosin on the cardiovascular and subjective effects of cocaine in a human laboratory study.

DETAILED DESCRIPTION:
Primary Objective: The primary objective is to determine the safety of treatment with doxazosin in cocaine-dependent volunteers by examining hemodynamic and subjective effects of administration of ascending doses of cocaine (0, 20mg, and 40mg) and a placebo dose during treatment with doxazosin.

Secondary Objectives: To evaluate the effect of doxazosin on the pharmacokinetics of intravenously administered cocaine; To determine effects of treatment with doxazosin, as compared to placebo, on subjective effects produced by administration of cocaine or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking volunteers who are not seeking treatment at the time of the study.
* Be between 18-55 years of age.
* Meet DSM-IV TR criteria for cocaine dependence; participants may or may not meet criteria for nicotine dependence. Nicotine dependence is allowed but not required because most cocaine users smoke cigarettes.
* Have a self-reported history of using cocaine by the smoked or IV route.
* Have vital signs as follows: supine blood pressure > 100/65 mm Hg, a seated blood pressure of > 90/60 mm Hg and < 150/90 mm Hg, and an orthostatic change < 20 mm Hg systolic or <10 mm Hg diastolic on standing. Resting pulse must be < 90 bpm.
* Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) within normal limits.
* Have a baseline EKG that demonstrates clinically normal sinus rhythm, clinically normal conduction, and no clinically significant arrhythmias.
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.

Exclusion Criteria:

* Meet DSM-IV TR criteria for dependence on drugs other than cocaine or nicotine.
* Have any history or evidence suggestive of seizure disorder or brain injury.
* Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, or epileptic seizure.
* Have neurological or psychiatric disorders, such as: psychosis, bipolar illness or major depression as assessed by MINI; organic brain disease or dementia assessed by clinical interview; history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of suicide attempts within the past year and/or current suicidal ideation/plan.
* Have evidence of clinically significant heart disease or hypertension, as determined by the PI.
* Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
* Have symptomatic HIV or are taking antiretroviral medication.
* Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation.
* Have asthma or currently use theophylline or other sympathomimetics.
* Have any other illness, condition, or use of psychotropic medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Criteria for Discontinuation Following Initiation:

Participants will be discharged if they have a positive breath test indicating use of alcohol or a urine test indicating illicit use of drugs while in the MED-VAMC, if they do not comply with study procedures, or if they do not tolerate the study drugs.

Subject Selection Criteria Rationale for Route of Administration:

Participants are required to have used cocaine by the IV or smoked route to avoid exposing participants to drugs by routes of administration that produce more intensive interoceptive effects than usually used by the participants. Prior experience with smoked cocaine is allowed (rather than restricting the population to those with experience with IV cocaine) because smoked cocaine reaches brain sites of action as rapidly as does intravenously administered cocaine and smoked cocaine produces effects that are comparable to IV cocaine. Speed of administration (and rate of delivery to brain) of stimulant drugs likely impacts subjective and cardiovascular effects, so smoked and intravenously administered cocaine produce similar subjective effects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The effects of treatment with doxazosin on cardiovascular effects after administration of ascending doses of cocaine (0, 20mg, and 40mg) and a placebo dose.
  Blood pressure (resting and orthostatic) will be assessed daily prior to dosing. Heart rate, EKG, and blood pressure will be recorded throughout and after experimental sessions using an automatic monitoring system. Participants will be monitored for stability on days 11 and 12 and discharged from the hospital on day 13.

SECONDARY OUTCOMES:
The effects of treatment with doxazosin, as compared to placebo, on subjective measures produced by administration of cocaine or placebo.
  Visual-analogue scale ratings of "any cocaine effect", "high", "good effects", "bad effects", "like cocaine", "desire cocaine", "depressed", "anxious", "stimulated", and "if you had access to cocaine right now, how likely would you be to use it?" will be collected at -15 min, 5 min, 10 min, 15 min, 20 min, 30 min, and 45 min after cocaine dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael Debakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Derived] Newton TF, De La Garza R 2nd, Brown G, Kosten TR, Mahoney JJ 3rd, Haile CN. Noradrenergic alpha(1) receptor antagonist treatment attenuates positive subjective effects of cocaine in humans: a randomized trial. PLoS One. 2012;7(2):e30854. doi: 10.1371/journal.pone.0030854. Epub 2012 Feb 3. PMID 22319592